CLINICAL TRIAL: NCT03306537
Title: A Quality Assurance Study of Respiratory Rate Measurements on Obese Patients With a Novel Monitoring Technology
Brief Title: Sensor Validation Study - Quality Assurance
Status: Completed | Type: Observational
Sponsor: PMD Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: PMD-CS-011
Record Dates: First submitted 2017-09-29; First posted 2017-10-11 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Respiratory Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: RespiraSense Respiratory Rate Monitor — RespiraSense device will be attached at the same time as the capnograph (gold standard) and both will measure simultaneously for one hour

SUMMARY:
The respiratory rate is an important parameter in clinical medicine. It is defined as the number of breaths per minute. Currently this is measured at the bedside in clinical practice by counting the breaths, however the gold standard for measuring this vital sign is the capnograph. For the patient, this involves wearing a tube in their nose and around their ears while trying to minimise their movement and talking so that the measurements can be taken.

A new respiratory rate monitor, RespiraSense, is non-invasive and measures the respiratory rate by measuring the displacement between the ribs and abdomen. This research study is intended to validate that this technology is effective and accurate on people with a bigger body mass.

Subjects with a BMI > 35 will be invited to participate should they meet all of the eligibility criteria. If patients agree to participate, following informed consent, subjects will be monitored for one hour with both the capnograph and RespiraSense measuring at the same time so their results can be compared

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 Years
* Have a BMI ≥35

  * For the sub-group analysis at least 5 subjects with a BMI 35-49 and at least 5 BMI > 50 will be needed
* Are willing to voluntarily sign a statement of informed consent to participate in this investigation

Exclusion Criteria:

* Allergic to medical grade skin adhesive
* Continuous oral long term steroid use. To be free from oral steroid use this is defined as not using oral steroids in the 4 weeks previous to enrolment
* Patients under the influence of substance abuse (drug or alcohol) that may interfere with their ability to cooperate and comply with the investigation procedures
* Any disorder, including cognitive dysfunction, which would affect the ability to accurately complete questionnaires and freely give full informed consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Obese patients with a BMI ≥35
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Comparison of PMD RespiraSense against capnography in obese patients. | 1 hour
  Analysed using a Bland Altman (BA) analysis to measure limits of agreement between both methods. The BA analysis will correct for repeated measures within each subject if required. In addition, a Deming Regression will be performed on the collected data.

SECONDARY OUTCOMES:
Comparison of PMD RespiraSense in obese patients with BMI below 50 and those with BMI of 50 or above. | 1 hour
  Analysed using a Bland Altman (BA) analysis to measure limits of agreement between both methods. The BA analysis will correct for repeated measures within each subject if required. In addition, a Deming Regression will be performed on the collected data.
Identification of any accuracy spread patterns as BMI increases. | 1 hour
  Analysed using a Bland Altman (BA) analysis to measure limits of agreement between both methods. The BA analysis will correct for repeated measures within each subject if required. In addition, a Deming Regression will be performed on the collected data.
Collection of feedback on device comfort when worn by patients with high BMI. | 1 hour
  Will not be analysed formally.

OTHER OUTCOMES:
Exploratory: To measure RespiraSense device alarm generation and assess the rationale behind these to determine if false alarms and therefore alarm fatigue is occurring | 1 hour
  Will not be analysed formally.

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Albon, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Queen Alexandra Hospital, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No